CLINICAL TRIAL: NCT02243657
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Multiple Oral Doses of ASP3652 in Healthy Young and Elderly Male and Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Effects in and on the Body of Healthy Young and Elderly Male and Female Subjects of Ascending Multiple Oral Doses of ASP3652
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3652-CL-0002; 2008-006416-38 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP3652; Pharmacodynamics of ASP3652
Keywords: ASP3652; Age; Gender; Pharmacokinetics; Pharmacodynamics; Phase 1; Multiple Ascending Doses (MAD)
MeSH Terms: conditions — Coitus | interventions — ASP3652

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1: Placebo dose level (Placebo Comparator)
  Interventions: Drug: Placebo
- 2: ASP3652 lowest dose level twice daily (Experimental)
  Interventions: Drug: ASP3652
- 3:ASP3652 low dose level twice daily (Experimental)
  Interventions: Drug: ASP3652
- 4: ASP3652 medium dose level twice daily (Experimental)
  Interventions: Drug: ASP3652
- 5: ASP3652 high dose level twice daily (Experimental)
  Interventions: Drug: ASP3652
- 6: ASP3652 highest dose level once daily (Experimental)
  Interventions: Drug: ASP3652

INTERVENTIONS:
Drug: ASP3652 — oral
  Arms: 2: ASP3652 lowest dose level twice daily; 3:ASP3652 low dose level twice daily; 4: ASP3652 medium dose level twice daily; 5: ASP3652 high dose level twice daily; 6: ASP3652 highest dose level once daily
Drug: Placebo — oral
  Arms: 1: Placebo dose level

SUMMARY:
The study investigates how safe ASP3652 is and how well it is tolerated when taken as multiple doses. The study also assesses how quickly and to what extent it is absorbed and eliminated from the body. In addition, the effects of age and gender are investigated.

The study consists of two parts. In Part 1 four dose levels are administered to four separate groups initially. Two additional dosages are then investigated. Subjects receive either a once-daily dose (QD) or twice-daily dose (BID) of ASP3652 or placebo.

Part 2 is performed in one group of elderly healthy male or female (post-menopausal) subjects. Subjects receive either a twice daily dose (BID) of ASP3652 or placebo.

For both parts of the study, the subjects stay in the clinic for one period of 18 days.

DETAILED DESCRIPTION:
This is a Multiple Ascending Dose (MAD) study with two parts. Screening for both parts takes place between Days -28 and -3. Subjects are admitted to the clinic on Day -2, and discharged on Day 16. They return for an End of Study Visit (ESV) between 7 and 14 days after (early) discharge.

Part 1 evaluates the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ASP3652 following ascending multiple oral doses. The initially planned four dose levels or matching placebo are given to four separate groups. Thereafter two additional dosage levels are further investigated. All groups receive a single dose of ASP3652 administered in the morning of Day 1 and Day 14, and twice-daily doses administered from Day 2 to Day 13 under fasted conditions, except the last group which receives all dosages once daily from Day 1 to Day 14.

Part 2 evaluates the safety, tolerability, PK and PD of ASP3652 following ascending multiple oral doses in healthy elderly male and female subjects. This part contains a single, placebo-controlled group. All subjects receive twice daily doses and administration is based on the results of Part 1.

All subjects in both parts receive training for Neurocognitive Test Battery (NTB) and tests for monitoring of psychotropic effects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5-30.0 kg/m2 for both male and female subjects.
* Male subject is non-fertile, i.e. surgically sterilized or practices an adequate contraceptive method to prevent pregnancies.
* Female subject is of non-child bearing potential, i.e. post menopausal, surgically sterilized, hysterectomy in medical history, or practices adequate (double barrier) non-hormonal contraceptive method to prevent pregnancies.

Exclusion Criteria:

* Pregnant or breast feeding within 6 months before screening assessment.
* Presence or history of any clinically significant psychiatric disorder such as mania, depression or schizophrenia.
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Nature, frequency and severity of adverse events | Screening to 14 days after discharge
Physical examination and vital signs | Screening to 14 days after discharge
Body temperature | Screening to 14 days after discharge
Routine safety laboratory tests | Screening to 14 days after discharge
12 -lead Electrocardiogram (ECG) | Screening to 14 days after discharge
Holter ECG | Day -1 and Day14
Monitoring of psychotropic / cannabinoids-like effects | Screening to 14 days after discharge
Neurocognition Test Battery (NTB) | Screening to 14 days after discharge
Examination for skin lesions | Screening to 14 days after discharge
Pharmacokinetic (PK) profile in plasma for first dose measured by area under the plasma concentration - time curve from time zero to infinity (AUCinf) | Day 1 to Day 2
PK profile in plasma for first dose measured by area under the plasma concentration - time curve from time zero to time of last measurable concentration (AUClast) | Day 1 to Day 2
PK profile in plasma for first dose measured by maximum plasma concentration (Cmax) | Day 1 to Day 2
PK profile in plasma for first dose measured by time to attain Cmax (tmax) | Day 1 to Day 2
PK profile in plasma for first dose measured by elimination half-life (t½) | Day 1 to Day 2
PK profile in plasma for first dose measured by absorption lag time (tlag) | Day 1 to Day 2
PK profile in plasma for first dose measured by apparent volume of distribution during the terminal phase (Vz/F) | Day 1 to Day 2
PK profile in plasma for first dose measured by apparent total clearance of the drug from plasma after oral administration (CL/F) | Day 1 to Day 2
PK profile in urine for first dose measured by cumulative amount of unchanged drug excreted into the urine from time zero to time of last measurable concentration (Aelast) | Day 1 to Day 2
PK profile in urine for first dose measured by cumulative amount of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf) | Day 1 to Day 2
PK profile in urine for first dose measured by percentage of unchanged drug excreted into the urine from time zero to time of last measurable concentration (Aelast%) | Day 1 to Day 2
PK profile in urine for first dose measured by percentage of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf%) | Day 1 to Day 2
PK profile in urine for first dose measured by renal clearance of the drug from plasma (CLR) | Day 1 to Day 2
PK profile in plasma for last dose measured by area under the plasma concentration - time curve between consecutive dosing (AUCtau) | Day 14 to Day 16
  Only for Bis in die (twice daily) (BID) dosing
PK profile in plasma for last dose measured by area under the plasma concentration- time curve from the time of dosing up to 24 hours (AUC0-24) | Day 14 to Day 16
  Only for BID dosing
PK profile in plasma for last dose measured by tmax | Day 14 to Day 16
PK profile in plasma for last dose measured by Cmax | Day 14 to Day 16
PK profile in plasma for last dose measured by t½ | Day 14 to Day 16
PK profile in plasma for last dose measured by Vz/F | Day 14 to Day 16
PK profile in plasma for last dose measured by CL/F | Day 14 to Day 16
PK profile in plasma for last dose measured by accumulation ratio (Rac) | Day 14 to Day 16
PK profile in plasma for last dose measured by Peak Trough Ratio (PTR) | Day 14 to Day 16
PK profile in plasma for last dose measured by plasma concentration at the end of a dosing interval at steady state (Ctrough) | Day 14 to Day 16
PK profile in urine for last dose measured by cumulative amount of drug excreted into urine over the time interval between consecutive dosing (Aetau) | Day 14 to Day 16
  Only for BID dosing
PK profile in urine for last dose measured by fraction of the drug excreted into urine (Aetau) over the time interval between consecutive dosing (Aetau%) | Day 14 to Day 16
  Only for BID dosing
PK profile in urine for last dose measured by CLR | Day 14 to Day 16
  Only for BID dosing
PK profile in urine for last dose measured by cumulative amount of unchanged drug excreted into the urine from 0 to 24 hours (Ae0-24) | Day 14 to Day 16
  Only for BID dosing
PK profile in urine for last dose measured by percentage of unchanged drug excreted into the urine from 0 to 24 hours (Ae0-24%) | Day 14 to Day 16

SECONDARY OUTCOMES:
Assessment of Pharmacodynamics measured by Ex vivo enzyme activity in mononuclear cells | Day -1 to Day 16
Pharmacodynamics measured by levels of arachidonoyl-ethanolamide (AEA) in plasma and seminal fluid (exploratory) | Day -2 or -1 and day 11, 12 or 13
Pharmacodynamics measured by levels of oleoyl-ethanolamide (OEA) in plasma and seminal fluid (exploratory) | Day -2 or -1 and day 11, 12 or 13
Pharmacodynamics measured by levels of palmitoyl-ethanolamide (PEA) in plasma and seminal fluid (exploratory) | Day -2 or -1 and day 11, 12 or 13
Assessment of Pharmacodynamics measured by intraocular pressure (IOP) (exploratory) | Day -1 to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- PRA International, Groningen, Netherlands